CLINICAL TRIAL: NCT06760741
Title: PREVENPANC Project: a Spanish Multicenter Study for Pancreatic Cancer Prevention
Acronym: PREVENPANC
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Hospital Universitario de Canarias (Other); Hospital Universitario Marqués de Valdecilla (Other); Hospital Universitario Ramon y Cajal (Other); Hospital de Cruces (Other); Hospital Universitario de Puerta de Hierro (Unknown); Clinica Universidad de Navarra, Universidad de Navarra (Other); Complexo Hospitalario de Ourense (Other)
Responsible Party: Principal Investigator, Irina Sofia Luzko Scheid, Principal Investigator. Gastroenterologist. Irina Luzko, Hospital Clinic of Barcelona
Other Study IDs: PREVENPANC
Record Dates: First submitted 2024-12-18; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Cancer, Adult; Hereditary Pancreatic Cancer; Familial Pancreatic Cancer
Keywords: Screening; Pancreatic cancer; High risk pancreatic cancer; Hereditary pancreatic cancer; Familial pancreatic cancer; miRNA pancreatic cancer
MeSH Terms: conditions — Pancreatic cancer, adult; Pancreatic carcinoma, familial; Pancreatic Neoplasms | interventions — Hematologic Tests; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Serum Plasma Pancreatic tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Population-based Pancreatic Cancer Cohort: PROSPECTIVE COHORT: Prospective inclusion of all patients from the general population diagnosed with pancreatic cancer over one year in each center.
  Interventions: Genetic: Multigene panel; Genetic: Generation of 3D Pancreatic Organoids
- Retrospective cohort: *RETROSPECTIVE COHORT: Enrollment of individuals from families with familial or hereditary pancreatic cancer who have been under follow-up since 2014 by the High Risk Digestive Cancer Clinic of the centers and who agree to participate in the study.
  Interventions: Diagnostic Test: Other; Diagnostic Test: miRNA measurement in blood
- Healthy control cohort: *HEALTHY CONTROLS: Enrolled from general gastroenterology consultations with imaging tests performed as part of routine clinical practice that rule out pancreatic pathology.

INTERVENTIONS:
Genetic: Multigene panel — Germline Genetic Testing: Germline genetic testing will be performed on all patients with pancreatic cancer (PC) using a custom multigene panel. This panel includes 25 candidate genetic variants of interest and 13 clinically recognized genes associated with a higher risk of PC.
  DNA Extraction: Germline DNA will be extracted from peripheral blood samples using the QIAamp DNA Blood Kit (Qiagen, Redwood City, CA, USA) following the manufacturer's instructions. The concentration of double-stranded DNA will be measured using a fluorometric method (Qubit, Thermo Fisher Scientific).
  Groups: Population-based Pancreatic Cancer Cohort
Diagnostic Test: Other — 1. Characterization of Suspected Pancreatic Cancer Lesions:
     Characterization of suspected pancreatic cancer (PC) lesions identified by endoscopic ultrasound (EUS) and/or magnetic resonance imaging (MRI) in patients undergoing screening since 2014. This includes lesion type (solid or cystic), rapid cyst growth exceeding 4 mm per year, location, size, potential assessment of resectability, lobulocentric parenchymal atrophy, and Wirsung duct dilation. Clinically relevant suspected lesions will be defined as solid lesions, intraductal papillary mucinous neoplasms (IPMN), cystic lesions ≥10 mm, and cystic lesions with mural nodules.
  2. Determination of CA 19-9 and Glycated Hemoglobin:
  Measurement of CA 19-9 levels and glycated hemoglobin (HbA1c) as part of the diagnostic and monitoring process.
  Other Names: RMN; Blood test; Ecoendoscopia biliopancreática
  Groups: Retrospective cohort
Diagnostic Test: miRNA measurement in blood — Analysis of miRNA Expression in plasma:
  The expression of circulating miRNAs (in plasma) will be analyzed using quantitative reverse transcription polymerase chain reaction (qRT-PCR). The signature includes two miRNAs (miR-33a-3p and miR-320a) combined with CA 19-9.
  Groups: Retrospective cohort
Genetic: Generation of 3D Pancreatic Organoids — Generation of 3D Pancreatic Organoids for Complementary Analyses:
  3D pancreatic organoids will be generated for complementary analyses involving in vitro functional studies to evaluate the pathogenicity of novel genes (selected based on the results of the multigene panel). These organoids will be developed from surgical samples obtained from five patients undergoing surgery as part of clinical care.
  Groups: Population-based Pancreatic Cancer Cohort

SUMMARY:
Background: Pancreatic cancer (PC) is an aggressive cancer with only a 7% 5-year survival rate, primarily due to late-stage diagnosis. In Spain, its incidence is rising, and by 2030, it is expected to become the second leading cause of cancer-related death worldwide. Approximately 3% of PCs occur in the context of hereditary pancreatic cancer (HPC) predisposition syndromes. Studies have shown that up to 40% of genetic mutations associated with PC in individuals under 60 years old would not have been identified using traditional clinical criteria for genetic testing. Presymptomatic genetic testing is recommended for relatives of patients with hereditary syndromes to identify those at higher risk of PC and to include them in screening programs to alter the natural history of the disease. However, there is no robust evidence supporting the best tool for early diagnosis in at-risk individuals. Currently, screening relies on endoscopic ultrasound or magnetic resonance imaging, which yield suboptimal results.

Aims: By studying the clinical, molecular, and genetic characteristics of PC patients and their families, this project aims to identify factors conferring higher PC risk and to adopt preventive measures while evaluating the efficacy of current screening strategies. Additionally, the project includes a traslational subproject to identify new hereditary genes associated with increased PC risk and novel molecules (biomarkers, specifically miRNAs) with diagnostic potential. These biomarkers could serve as non-invasive tools to identify individuals at increased risk of PC through blood tests, enabling preventive measures or early diagnosis.

Given the low incidence of PC (albeit with high mortality), collaborative studies are essential to achieve meaningful results. The current project represents the first Spanish multicenter population-based registry for PC, integrating clinical data and biological sample collection alongside a control group. Its goal is to prevent PC and foster collaboration between basic research and clinical application in Spain within a proven collaborative framework.

Establishing the best strategy to detect high-risk individuals for PC within the general population.

Identifying new PC risk genes to expand the identification of at-risk individuals.

Determining effective prevention strategies for high-risk individuals. Creating a national network, "PREVENPANC," for collaborative PC research, including the collection of biological samples (blood) from all enrolled patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a recent diagnosis of pancreatic cancer in the general population.
* High-risk individuals under follow-up in high-risk clinics (hereditary syndromes, familial pancreatic cancer).

Exclusion Criteria:

* Patients under 18 years old.
* Patients who have undergone treatment for pancreatic cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Population-Based Cohort:
     Prospective inclusion of all patients diagnosed with pancreatic cancer (PC) over a 12-month period at participating centers, paired with a control group of individuals without known pancreatic pathology. Controls will be matched by age, sex, and self-identified gender.
  2. Retrospective Cohort (Individuals from Families with Familial Pancreatic Cancer or Hereditary Pancreatic Cancer):
  Observational multicenter study with retrospective inclusion of all individuals from families with familial pancreatic cancer (FPC) or hereditary pancreatic cancer (HPC) who have been under follow-up from 2014 to the present in the High Risk Digestive Cancer Clinics of the participating centers. Peripheral blood samples (serum, plasma, and DNA) from most of these individuals are currently available in biobank storage.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Identification of Pancreatic Cancer Risk Groups within the General Population | Until March 2026
  *Clinical Protocol:
  - Identify the factors and risk groups globally associated with pancreatic cancer (PC).
Identification of Pancreatic Cancer Risk Groups within the General Population | Until March 2026
  *Clinical Protocol:
  - Determine the prevalence of germline genetic mutations in individuals diagnosed with PC within the population-based cohort over one year.
Identification of Pancreatic Cancer Risk Groups within the General Population | Until March 2026
  *Translational Protocol:
  - Discover and validate new hereditary genes associated with an increased risk of PC through targeted sequencing using a multigene panel.
Evaluate Screening Strategies in High-Risk Individuals | Until October 2026
  *Clinical Protocol:
  -Identify specific risk factors associated with pancreatic cancer (PC) in families with familial pancreatic cancer (FPC) or hereditary pancreatic cancer (HPC).
Evaluate Screening Strategies in High-Risk Individuals | Until October 2026
  *Clinical Protocol:
  -Determine the prevalence of PC in families diagnosed with FPC and HPC in our setting.
Evaluate Screening Strategies in High-Risk Individuals | Until October 2026
  *Clinical Protocol:
  - Assess the efficacy of PC screening strategies in these high-risk groups (FPC and HPC).
Evaluate Screening Strategies in High-Risk Individuals | Until October 2026
  *Translational Protocol:
  -Evaluate the non-invasive diagnostic yield of selected mentioned miRNAs as biomarkers for PC screening and early diagnosis in FPC and HPC groups using qRT-PCR.

SECONDARY OUTCOMES:
Identification of Pancreatic Cancer Risk Groups within the General Population | Until March 2026
  *Clinical Protocol:
  - Establish the most effective strategy for identifying individuals with a hereditary predisposition to PC.
Identification of Pancreatic Cancer Risk Groups within the General Population | Until March 2026
  *Translational Protocol:
  - Evaluate the pathogenicity of identified genetic variants through in vitro functional studies using the generation and modification of 3D pancreatic organoids.

OTHER OUTCOMES:
Establish a Spanish Multicenter Network for Collaborative Research on Pancreatic Cancer Prevention in Our Setting ("PREVENPANC") | November 2025
  Create a Cohort with Clinical Information and Biological Samples:
  Establish a cohort comprising individuals with and without pancreatic pathology as a control group for future projects within the PREVENPANC network.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Llach J, Luzko I, Earl J, Barreto E, Rodriguez-Garrote M, Lleixa M, Herrera-Pariente C, Fernandez G, Munoz J, Bonjoch L, Sauri T, Ausania F, Ocana T, Moreno L, Grau E, Oriola J, Alvarez-Mora MI, Herreros-Villanueva M, Castellvi-Bel S, Balaguer F, Bujanda L, Moreira L. Should We Offer Universal Germline Genetic Testing to All Patients with Pancreatic Cancer? A Multicenter Study. Cancers (Basel). 2024 Nov 9;16(22):3779. doi: 10.3390/cancers16223779. PMID 39594734
- [Background] Vila-Navarro E, Duran-Sanchon S, Vila-Casadesus M, Moreira L, Gines A, Cuatrecasas M, Lozano JJ, Bujanda L, Castells A, Gironella M. Novel Circulating miRNA Signatures for Early Detection of Pancreatic Neoplasia. Clin Transl Gastroenterol. 2019 Apr;10(4):e00029. doi: 10.14309/ctg.0000000000000029. PMID 31009404